CLINICAL TRIAL: NCT03724123
Title: Machine Learning-Based Risk Profile Classification of Patients Undergoing Elective Heart Valve Surgery
Status: Completed | Type: Observational
Sponsor: Kepler University Hospital (Other)
Collaborators: Institute of Bioinformatics, JKU Linz (Unknown)
Responsible Party: Principal Investigator, Jens Meier, Prof. Dr., Kepler University Hospital
Other Study IDs: K-82-15
Record Dates: First submitted 2018-10-25; First posted 2018-10-30 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Heart Valve Diseases; Surgery--Complications
Keywords: random forests; heart valve surgery; support vector machines; artificial neural networks
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Machine learning methods potentially provide a highly accurate and detailed assessment of expected individual patient risk before elective cardiac surgery. Correct anticipation of this risk allows for improved counseling of patients and avoidance of possible complications. The investigators therefore investigate the benefit of modern machine learning methods in personalized risk prediction in patients undergoing elective heart valve surgery.

DETAILED DESCRIPTION:
The investigators performe a monocentric retrospective study in patients who underwent elective heart valve surgery between January 1, 2008, and December 31, 2014 at our center. The investigators use random forests, artificial neural networks, and support vector machines to predict the 30-days mortality from a subset of demographic and preoperative parameters. Exclusion criteria were re-operation of the same patient, patients that needed anterograde cerebral perfusion due to aortic arch surgery, and patients with grown up congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent heart valve surgery of any kind between 2008-01-01 and 2014-12-31 were included.

Exclusion Criteria:

* re-operation of the same patient
* patients that needed anterograde cerebral perfusion due to aortic arch surgery
* patients with grown-up congenital heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent heart valve surgery of any kind between 2008-01-01 and 2014-12-31 were included.
Sampling Method: Non-Probability Sample
Enrollment: 2229 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Area under the curve for different prediction models | Patients will included from 01.01.2008 - 31.12.2014
  Three different predictions models will be used.

REFERENCES:
- [Derived] Bodenhofer U, Haslinger-Eisterer B, Minichmayer A, Hermanutz G, Meier J. Machine learning-based risk profile classification of patients undergoing elective heart valve surgery. Eur J Cardiothorac Surg. 2021 Dec 1;60(6):1378-1385. doi: 10.1093/ejcts/ezab219. PMID 34050368